CLINICAL TRIAL: NCT03981874
Title: Comparative Study of Peripheral Facial Paralysis Sequelae Based on the Initial Medical Care of Lyme Disease Among Children
Brief Title: Peripheral Facial Paralysis Sequelae in Lyme Disease Among Children
Acronym: LYMEPED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P/2019/419
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Lyme Disease
Keywords: neuroborreliosis; facial palsy; children
MeSH Terms: conditions — Lyme Disease; Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telephonic interview (Experimental): Parents or patients will be contacted by phone in order to precise whether there are persistent sequelae or not
  Interventions: Other: telephonic interview

INTERVENTIONS:
Other: telephonic interview — Telephonic interview

SUMMARY:
Neuroborreliosis (NB) is the second most frequent manifestation of Lyme disease. Painful meningoradiculitis is the most common neurologic manifestation in adults while facial nerve palsy (FP) and lymphocytic meningitis is predominant in children. FP is a common reason for pediatric consultation and FP due to Lyme borreliosis (LB) represents about 50% of the child's FP in an endemic area.

The action to be taken is not formally defined for a child consulting for FP in a Lyme disease endemic area.

The new recommendations of the High Authority of Health of June 2018 recommend to carry out a blood serology in first intention, in search of a NB in a child consulting for a peripheral facial paralysis. If this is positive, a lumbar puncture will be performed in search of meningitis. In the case of negative serology, a close clinical surveillance and sometimes serological control is necessary, in order to reassess the diagnosis. In adult recommendations, a lumbar puncture is performed first in any patient consulting for facial paralysis in LB endemic area.

The main objective of this study was to describe the clinical and biological characteristics of pediatric NB with FP. Others objectives were to describe the diagnostic and therapeutic behavior of a child consulting at university hospital for a facial nerve palsy, to compare the initial gravity of facial nerve palsy, the duration of the paralysis and sequels depending on the diagnosis and treatment initiated.

ELIGIBILITY:
Inclusion Criteria:

* Children consulting for peripheral facial palsy

Exclusion Criteria:

* Children consulting for central facial palsy
* Children with congenital peripheral facial palsy
* Children with surgery and trauma in the area of the facial nerve,
* Children with peripheral facial palsy with previous diagnosis
* Children whose parents refuse the study participation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-07-29 (Estimated); Study Completion 2019-07-29 (Estimated)

PRIMARY OUTCOMES:
Assesment of persistent sequelae | 4 years
  Facial paralysis duration assesment and persistence of physical sequelae at time of the telephonic call using House & Brackmann classification for facial function.
  This grading system has 6 levels, used for middle- to long-term monitoring:
  I. Normal II. Mild dysfunction III. Moderate dysfunction IV. Moderately severe dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Anxionnat, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No